CLINICAL TRIAL: NCT00666874
Title: Effect of Weight Loss and Lifestyle Changes on Vascular Inflammatory Markers in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Dario Giugliano, MD, Department of Geriatrics and Metabolic Diseases, Second University of Naples
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGGM/02/1999
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
Keywords: Obesity, lifestyle, vascular inflammation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Detailed advice about how to achieve a reduction of weight of 10% or more through a low-energy Mediterranean-style diet and increased physical activity.
  Interventions: Behavioral: lifestyle changes
- 2 (Active Comparator): General information about healthy food choices and exercise
  Interventions: Behavioral: Control - general information

INTERVENTIONS:
Behavioral: lifestyle changes — Detailed advice about how to achieve a reduction of weight of 10% or more through a low-energy Mediterranean-style diet and increased physical activity.
  Other Names: lifestyle
  Arms: 1
Behavioral: Control - general information — General information about healthy food choices and exercise
  Other Names: control
  Arms: 2

SUMMARY:
Obesity is an independent risk factor for cardiovascular disease, which may be mediated by increased secretion of proinflammatory cytokines by adipose tissue.

To determine the effect of a program of changes in lifestyle designed to obtain a sustained reduction of body weight on markers of systemic vascular inflammation and insulin resistance.

Randomized single-blind trial conducted from February 1999 to February 2002 at a university hospital in Italy.

One hundred twenty premenopausal obese women (body mass index 30) aged 20 to 46 years without diabetes, hypertension, or hyperlipidemia.

The 60 women randomly assigned to the intervention group received detailed advice about how to achieve a reduction of weight of 10% or more through a low-energy Mediterranean-style diet and increased physical activity. The control group (n = 60) was given general information about healthy food choices and exercise.

ELIGIBILITY:
Inclusion Criteria:

* obese premenopausal women,
* aged 20 to 46 years
* sedentary (<1 h/wk of physical activity)
* with no evidence of participation in diet reduction programs within the last 6 months.

Exclusion Criteria:

* type 2 diabetes mellitus or impaired glucose tolerance (plasma glucose levels of 140-200 mg/dL [7.8-11.1 mmol/L] 2 hours after a 75-g oral glucose load)
* hypertension (blood pressure >140/90 mm Hg)
* cardiovascular disease, psychiatric problems
* history of alcohol abuse (intake of 500 g/wk in the last year)
* current smoking
* any medication use.

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 1999-02; Primary Completion 2001-12 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Vascular inflammatory markers (IL-6, IL-18, CRP, Adiponectin) | 24 months

SECONDARY OUTCOMES:
Insulin resistance (HOMA) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD,PhD, Principal Investigator — Department of Geriatrics and metabolic Diseases
Locations (1):
- Department of Geriatrics and Metabolic Diseases, Naples, Italy

REFERENCES:
- [Result] Esposito K, Pontillo A, Di Palo C, Giugliano G, Masella M, Marfella R, Giugliano D. Effect of weight loss and lifestyle changes on vascular inflammatory markers in obese women: a randomized trial. JAMA. 2003 Apr 9;289(14):1799-804. doi: 10.1001/jama.289.14.1799. PMID 12684358